CLINICAL TRIAL: NCT06963918
Title: Effect of Expiratory Muscle Strength Training on Forward Trunk Flexion in Parkinson's Disease
Brief Title: Expiratory Muscle Training and Trunk Flexion in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Kateřina Dvořáková, Physiotherapist, General University Hospital, Prague
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17/25 S-IV
Record Dates: First submitted 2025-04-23; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Expiratory Muscle Strength Training; Forward Trunk Flexion
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Expiratory Muscle Strength Training (Experimental): The experimental group will first undergo a 4-week wait-to-start period, then participate in a 4-week expiratory muscle strength training program, followed by a 4-week follow-up phase.
  Interventions: Device: Expiratory muscle strength training

INTERVENTIONS:
Device: Expiratory muscle strength training — After the 4-week wait-to-start period during which they will not receive any intervention, will participants undergo a 4-week respiratory training program using the EMST150™ device (Expiratory Muscle Strength Trainer). EMST therapy sessions will be completed at home on 5 days (of the patients choosing) per week, performing five sets of five forceful exhalations through the EMST150™. The resistance of the device will be set to 75% of the patient's individual maximum expiratory pressure (MEP). The daily training will take approximately 15 minutes. Following the training period, patients will be observed for an additional 4 weeks to assess the sustainability of the potential training effects.

SUMMARY:
Postural abnormalities involving the trunk are prevalent in over 20% of patients with Parkinson's disease (PD). Pathological forward trunk flexion (FTF) is a drug-refractory complication in patients with PD leading to imbalance, pain and fall-related injuries. Deep abdominal muscle training is a key rehabilitation strategy for FTF, as muscles like the transversus abdominis and multifidus are crucial for lumbar stabilization. This training has been shown to improve body position and lumbar proprioception.

Abdominal muscles are also responsible for forced expiration. Expiratory muscle strength training (EMST) utilizing forced expiration through expiratory trainer has emerged as a beneficial intervention in the non-pharmacological management of PD, positively impacting clinical aspects such as dysphagia, dystussia, hypokinetic dysarthria, and drooling. EMG study showed large abdominal muscles activity, particularly the transversus abdominis and internus obliquus abdominis during EMST. Therefore, EMST might also be effective in improving lumbar stabilization.

Given the established role of abdominal muscles in trunk stabilization, it is plausible that activation of deep abdominal muscles during EMST with the right level of resistance might improve FTF in PD patients. No studies have yet examined the effect of EMST on posture in PD.

The primary aim of this study will be to evaluate the effect of EMST on forward trunk flexion in patients with Parkinson's disease.

The secondary aim will be to assess the potential duration of the EMST effect on postural abnormalities and its impact on patient stability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease
* Age ≥ 18 years
* MoCA (Montreal Cognitive Assessment) score ≥19
* Pathological forward trunk flexion defined as thoracic (≥25°) or lumbar (>15°) flexion during standing and walking, which completely disappears in the supine position.

Exclusion Criteria:

* Severe dyskinesia or "on-off" fluctuations
* Change in the PD medication in the last 3 months prior to enrollment
* History of major spinal surgery or musculoskeletal spinal disorders
* Need for assistive devices when rising from a chair or bed
* Other neurological, orthopedic, or cardiovascular comorbidities that could affect postural control
* Inadequate lip seal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in the forward trunk flexion (FTF) angle | Week 0, Week 8, Week 12
  Forward trunk flexion will be assessed using standardized postural photographs. Images will be taken with a camera mounted on a tripod positioned 1 meter above the ground and 3 meters from the participant. The participant will stand in tight-fitting clothing at a predefined location in front of a white wall with a calibration pattern. All camera parameters will remain unchanged throughout the study. Photographs will be analyzed using a semi-automated method, and the extent of forward trunk flexion will be classified according to standardized guidelines for axial postural abnormalities in Parkinson's disease.

SECONDARY OUTCOMES:
MDS-Unified Parkinson's Disease Rating Scale: Part II. and III. | Week 0, week 4, week 8, week 12
  This portion of the scale assesses the motor signs of Parkinson´s disease.The maximum total UPDRS score is 272, indicating the worst possible disability from Parkinson's Disease. The minimum total score is 0, indicating no disability from PD. Improvement greater than (-4.9) points or worsening more than (+4.2) points on MDS-UPDRS II+III represent a minimal clinically important difference.
Mini-Balance Evaluation Systems Test (Mini-BESTest) | Week 0, week 4, week 8, week 12
  The Mini-BESTest is a comprehensive clinical tool designed to assess balance and postural control. The test consists of 14 tasks, comprising a total of 28 items, each rated from 0 to 2, where 0 indicates severe impairment, 1 indicates moderate impairment and 2 stands for normal performance.
Pain Intensity - Numeric Rating Scale | Week 0, week 4, week 8, week 12
  Self-reported pain intensity on an 11-point scale (0 = no pain, 10 = worst imaginable pain).
The Parkinson's Disease Questionnaire (PDQ-39) | Week 0, week 4, week 8, week 12
  The 8-item questionnaire assesses quality of life in people with PD. The minimum score is 0, while the maximum is 100. A higher score indicates a lower quality of life.
Number of Falls in the Previous Month | Week 0, week 4, week 8, week 12
  Self-reported number of falls experienced in the preceding month.
Forced expiratory volume (FEV1) | Week 0, week 4, week 8, week 12.
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.
Forced vital capacity (FVC) | Week 0, week 4, week 8, week 12.
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.
Peak expiratory flow (PEF) | Week 0, week 4, week 8, week 12.
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chino K, Ohya T, Suzuki Y. Association between expiratory mouth pressure and abdominal muscle activity in healthy young males. Eur J Appl Physiol. 2024 Jul;124(7):2139-2151. doi: 10.1007/s00421-024-05430-5. Epub 2024 Mar 1. PMID 38427101
- [Background] Puntumetakul R, Chalermsan R, Hlaing SS, Tapanya W, Saiklang P, Boucaut R. The effect of core stabilization exercise on lumbar joint position sense in patients with subacute non-specific low back pain: a randomized controlled trial. J Phys Ther Sci. 2018 Nov;30(11):1390-1395. doi: 10.1589/jpts.30.1390. Epub 2018 Nov 6. PMID 30464372
- [Background] Hlaing SS, Puntumetakul R, Khine EE, Boucaut R. Effects of core stabilization exercise and strengthening exercise on proprioception, balance, muscle thickness and pain related outcomes in patients with subacute nonspecific low back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2021 Nov 30;22(1):998. doi: 10.1186/s12891-021-04858-6. PMID 34847915
- [Background] Szczygiel E, Blaut J, Zielonka-Pycka K, Tomaszewski K, Golec J, Czechowska D, Maslon A, Golec E. The Impact of Deep Muscle Training on the Quality of Posture and Breathing. J Mot Behav. 2018 Mar-Apr;50(2):219-227. doi: 10.1080/00222895.2017.1327413. Epub 2017 Aug 18. PMID 28820662
- [Background] Gandolfi M, Geroin C, Imbalzano G, Camozzi S, Menaspa Z, Tinazzi M, Alberto Artusi C. Treatment of axial postural abnormalities in parkinsonism disorders: A systematic review of pharmacological, rehabilitative and surgical interventions. Clin Park Relat Disord. 2024 Mar 12;10:100240. doi: 10.1016/j.prdoa.2024.100240. eCollection 2024. PMID 38596537
- [Background] Artusi CA, Geroin C, Imbalzano G, Camozzi S, Aldegheri S, Lopiano L, Tinazzi M, Bombieri N. Assessment of Axial Postural Abnormalities in Parkinsonism: Automatic Picture Analysis Software. Mov Disord Clin Pract. 2023 Feb 20;10(4):636-645. doi: 10.1002/mdc3.13692. eCollection 2023 Apr. PMID 37070056